CLINICAL TRIAL: NCT06747754
Title: Database HIV (DBHIV)-Costituzione di un Database di Pazienti HIV.
Brief Title: HIV Database (DBHIV)-Establishment of a Database of HIV Patients
Acronym: HIVDB
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID6741
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Database Management Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Establishment of a Database of HIV Patients — Establishment of a database that allows for systematic and continuous collection of data relating to clinical, laboratory and treatment characteristics of patients with HIV-1 for research purposes.
  Other Names: Database

SUMMARY:
In Italy, there are over 90,000 patients with HIV-1 infection on antiretroviral therapy (ART). The availability of different classes of antiretroviral drugs (nucleoside and non-nucleoside reverse transcriptase inhibitors (NRTIs, NNRTIs), protease inhibitors (PIs), integrase inhibitors (INSTIs) and viral entry inhibitors (IEs) that act in different phases of the HIV life cycle, together with careful patient management, has allowed us to obtain long-lasting therapeutic efficacy in the vast majority of Italian patients, making this infection a chronic disease.The introduction of combination antiretroviral therapy (cART) has completely revolutionized the management of HIV-positive patients, drastically reducing HIV-associated mortality and morbidity. In fact, the course of HIV infection has transformed into a chronic disease, and the number of HIV-infected patients over 50 years of age has increased significantly and the number of elderly subjects is progressively increasing. Furthermore, HIV infection seems to accelerate the aging process, causing immune system dysfunction, excess oxidative stress and increased inflammatory processes (inflammaging).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with chronic HIV infection (certified by a positive test for the detection of anti-HIV antibodies)
* Ability to sign the informed consent or signature of the declaration in lieu of consent in the case of deceased patients

Exclusion Criteria:

* lack of willingness to provide free and informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with HIV infection
Sampling Method: Non-Probability Sample
Enrollment: 4900 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishment of a database | 5 years
  Establishment of a database that allows for systematic and continuous collection of data relating to clinical, laboratory and treatment characteristics of patients with HIV-1 for research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Torti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Malattie Infettive, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No